CLINICAL TRIAL: NCT00661804
Title: A Longitudinal Cohort Study of Patients With Thalassemia in the Thalassemia Clinical Research Network
Brief Title: Evaluating People With Thalassemia: The Thalassemia Longitudinal Cohort (TLC) Study
Status: Completed | Type: Observational
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Thalassemia Clinical Research Network (Network)
Responsible Party: National Heart, Lung and Blood Institute, National Institutes of Health
Other Study IDs: 568; U01HL065238 (NIH)
Record Dates: First submitted 2008-04-16; First posted 2008-04-18 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-06

CONDITIONS: Thalassemia
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA and frozen plasma genetic biorepository
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Thalassemia cohort: Thalassemia as documented by clinical diagnosis, including:
  thalassemia (intermedia or major); HbH disease; HbH with non-deletional mutations, e.g., HbH Constant Spring E beta-thalassemia; Homozygous alpha-thalassemia (i.e., 4-gene alpha deletion or equivalent null alpha mutation); Other thalassemic conditions not explicitly excluded; Thalassemia intermedia due to heterozygous beta mutation with alpha-gene excess.
- Successful SCT cohort: Individuals who have received a successful hematopoietic SCT, defined as engraftment of all three cell lines and transfusion independence by 100 days post-transplant, for any of the disorders listed above;Monitored for end-organ injury related to thalassemia prior to their successful SCT;Participants who were enrolled in TCRN Registry or had a successful SCT after 01 Jan 2002.

SUMMARY:
Thalassemias are inherited blood disorders that can cause anemia and other health problems. The goal of this study is to collect information on complications of the disease among people who currently have or previously had thalassemia.

DETAILED DESCRIPTION:
Thalassemias are inherited blood disorders that are characterized by low levels of hemoglobin and healthy red blood cells. The two major types of thalassemia are alpha thalassemia and beta thalassemia, and there are several forms of each type. Symptoms can range from mild to severe and may include anemia, delayed growth, bone problems, and an enlarged spleen. People with mild forms of the disease may not need any treatment, while people with moderate to severe thalassemia may be treated with blood transfusions to refresh the healthy red blood cell supply, iron chelation therapy to remove excess iron from the body, and folic acid supplements to help build healthy red blood cells. Stem cell transplants can cure the disease, but they are not widely used because of the difficulty of finding donors. This study will establish a database of people with thalassemia and people who used to have thalassemia to examine the prevalence and incidence of complications related to the disease. Participants' DNA will be analyzed and plasma will be collected for use in future studies. Participants in this study may also be asked if they are interested in enrolling in other Thalassemia Clinical Research Network studies.

This study has enrolled people with thalassemia or people whose thalassemia was cured after undergoing a stem cell transplant. At a baseline study visit, participants with thalassemia will undergo a medical history interview; a medical record review; blood collection; and questionnaires on quality of life, nutritional status, and medication adherence. Follow-up visits will occur once a year for at least 3 years or for the duration of the study and will include repeat baseline testing. Participants who have undergone a successful stem cell transplant will attend only one study visit that will include a medical history interview, a medical record review, and quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria for People with Thalassemia:

* Thalassemia, as documented by clinical diagnosis, including the following types:

  1. Beta-thalassemia (intermedia or major)
  2. Hemoglobin H (HbH) disease
  3. HbH with non-deletional mutations (e.g., HbH Constant Spring)
  4. E-beta-thalassemia
  5. Homozygous alpha-thalassemia (i.e., 4-gene alpha deletion or equivalent null alpha mutation)
  6. Other thalassemic conditions not explicitly excluded
  7. Thalassemia intermedia due to heterozygous beta mutation with alpha-gene excess
* Requires at least annual monitoring for end-organ injury related to thalassemia, including all clinical measures specified in this study

Inclusion Criteria for People who Have Received a Successful Stem Cell Transplant:

* Received a successful hematopoietic stem cell transplant, defined as engraftment of all three cell lines and transfusion independence by 100 days post-transplant, for any of the thalassemia disorders listed above
* Monitored for end-organ injury related to thalassemia before their successful stem cell transplant, including all clinical measures specified in this study

Exclusion Criteria for People with Thalassemia:

* Has any of the following mild or mixed diagnoses:

  1. Thalassemia trait (i.e., single recessive beta-gene mutation, two-gene alpha-gene mutation)
  2. Thalassemia/Hb S, C, or D compound heterozygotes
  3. HbH with steady state hemoglobin above 9.0 g/dL and no history of significant thalassemia complications (e.g., endocrinopathies, cardiac dysfunction, growth impairment, pulmonary hypertension)
* Unable or unwilling to be followed annually

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients with thalassemia, as documented by clinical diagnosis, seen at sites funded by the Thalassemia Clinical Research Network (TCRN) and their satellites.
Sampling Method: Non-Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2007-05; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The prevalence and incidence of complications specific to thalassemia and its treatment among participants | Measured throughout the duration of the study

SECONDARY OUTCOMES:
Fertility and pregnancy outcomes; causes of mortality and changes in mortality risk; genotypic and phenotypic variation; and body iron burden | Measured throughout the duration of the study
Relationships among adherence, quality of life, and complications of thalassemia | Measured throughout the duration of the study

CONTACTS AND LOCATIONS:
Overall Officials: Ellis Neufeld, MD, PhD, Study Chair — Boston Children's Hospital; Janet Kwiatkowski, MD, Study Chair — Children's Hospital of Philadelphia
Locations (14):
- United States (10):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital of Oakland, Oakland, California
  - Stanford Hospital, Stanford, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Children's Memorial Hospital Chicago, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - Weill Medical College of Cornell University, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Southwestern Medical Center at Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
- Canada (3):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - Toronto Sick Kids, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
- Royal Free and University College London Medical School, London, England, United Kingdom

REFERENCES:
- [Derived] Trachtenberg FL, Mednick L, Kwiatkowski JL, Neufeld EJ, Haines D, Pakbaz Z, Thompson AA, Quinn CT, Grady R, Sobota A, Olivieri N, Horne R, Yamashita R; Thalassemia Clinical Research Network. Beliefs about chelation among thalassemia patients. Health Qual Life Outcomes. 2012 Dec 7;10:148. doi: 10.1186/1477-7525-10-148. PMID 23216870
- [Derived] Morris CR, Kim HY, Trachtenberg F, Wood J, Quinn CT, Sweeters N, Kwiatkowski JL, Thompson AA, Giardina PJ, Boudreaux J, Olivieri NF, Porter JB, Neufeld EJ, Vichinsky EP; Thalassemia Clinical Research Network. Risk factors and mortality associated with an elevated tricuspid regurgitant jet velocity measured by Doppler-echocardiography in thalassemia: a Thalassemia Clinical Research Network report. Blood. 2011 Oct 6;118(14):3794-802. doi: 10.1182/blood-2010-11-319152. Epub 2011 Jul 19. PMID 21772051